CLINICAL TRIAL: NCT05897619
Title: Pilot Trial Assessing Feasibility and Acceptability of a Novel Cognitive Behavioral Skills Mobile App for a Perinatal Population
Brief Title: Feasibility and Acceptability of a Novel Cognitive Behavioral Skills Mobile App for Pregnant and Postpartum Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-10025299
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Perinatal Anxiety; Perinatal Depression
Keywords: Perinatal; Pregnancy; Postpartum; Perinatal Mood and Anxiety Disorders; Cognitive Behavioral Therapy; Mobile App; mobile Health (mHealth)
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is an open pilot trial designed to assess the feasibility and acceptability of the Maya Perinatal Cognitive Behavioral Therapy Skills app. All participants will receive the same intervention and provide qualitative and quantitative feedback on app use and experience to inform future iterations of the app.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maya Perinatal Cognitive Behavioral Skills App (Experimental): Participants receive the Maya Perinatal Cognitive Behavioral Skills App for 6 weeks.
  Interventions: Behavioral: Experimental: Maya Perinatal Cognitive Behavioral Skills App

INTERVENTIONS:
Behavioral: Experimental: Maya Perinatal Cognitive Behavioral Skills App — The intervention includes the completion of a mobile skills app teaching evidence-based strategies tailored for perinatal mood and anxiety. Modules include psychoeducation, skill information, practice exercises, and homework.

SUMMARY:
This study aims to assess the feasibility and acceptability of the Maya Perinatal Cognitive Behavioral Skills App, a novel app for pregnant and postpartum individuals experiencing difficulties with mood, anxiety, or stress. Participants will complete the 12-module app to learn evidence-based strategies previously shown to help manage mood and anxiety. Assessments will include app feedback questionnaires, feedback interviews, a daily symptom tracker, and symptom measures. The study investigators hypothesizes that participants will find content to be helpful in developing skills to manage anxiety and mood difficulties during the perinatal period, and that the app interface, session structure, and pacing will be acceptable and feasible for this population. It is further hypothesized that increased Maya Perinatal Cognitive Behavioral Skills App use, engagement, and satisfaction will be associated with lower self-reported anxiety and mood symptoms.

DETAILED DESCRIPTION:
Individuals who are pregnant or postpartum are at a high risk of anxiety and mood difficulties. This has been linked to negative effects on the individual, developing baby (both in the womb and after birth), and family system. Despite this, there are significant barriers to getting mental health support while pregnant or as a new parent, particularly for those in disadvantaged communities. This study seeks to assess the feasibility and acceptability of a novel mobile health app among individuals who are pregnant or postpartum. The Maya Perinatal Cognitive Behavioral Skills App has been adapted from a previously studied Maya Cognitive Behavioral Skills App to specifically address the unique experiences of the perinatal population. The app includes 12 skill-based sessions using principles from cognitive behavioral therapy, an evidence-based treatment that can effectively address anxiety and mood symptoms. The app will be tested by pregnant and postpartum individuals, who will provide feedback on feasibility and acceptability. Participants will also complete screening measures assessing anxiety, mood, and trauma, which will be examined in the context of app use and engagement. Participants will be recruited from a range of settings in hopes of capturing a diverse sample in terms of race, cultural background, and financial means. Results will be used to inform future versions of the app to better suit this population.

ELIGIBILITY:
Inclusion Criteria:

* Female, Trans-male, non-binary, gender expansive, or gender questioning gestational carriers of pregnancy
* Currently pregnant or up to 12 months postpartum
* 18 years or older
* English proficiency
* Have access to a smartphone or other mobile device capable of receiving Short Message Service (SMS) pushes and complete Qualtrics surveys and App modules
* Be available to speak by phone or secure video-conference platform at points throughout the study.

Exclusion Criteria:

* Safety concerns at the time of enrollment, including, but not limited to, a response >0 on the EPDS question 10 or reported suicidal or self-harm thoughts or behaviors within one year of enrollment
* Current substance use disorder
* History of a bipolar or psychotic disorder, or current symptoms of psychosis or mania.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
User Version of the Mobile Application Rating Scale (uMARS) at midpoint | Midpoint (approximately 3 weeks)
  The uMARS is a 27-item self-report questionnaire assessing engagement, functionality, aesthetics, information, subjective quality, and perceived impact of an app. Total scores are calculated by averaging the items together, representing an overall perceived app quality score ranging from 1 (inadequate) to 5 (excellent).
User Version of the Mobile Application Rating Scale (uMARS) at post-intervention | Post-intervention (approximately 6 weeks)
  The uMARS is a 27-item self-report questionnaire assessing engagement, functionality, aesthetics, information, subjective quality, and perceived impact of an app. Total scores are calculated by averaging the items together, representing an overall perceived app quality score ranging from 1 (inadequate) to 5 (excellent).
User Version of the Mobile Application Rating Scale (uMARS) at follow-up | Follow-up (approximately 12 weeks)
  The uMARS is a 27-item self-report questionnaire assessing engagement, functionality, aesthetics, information, subjective quality, and perceived impact of an app. Total scores are calculated by averaging the items together, representing an overall perceived app quality score ranging from 1 (inadequate) to 5 (excellent).
Quantitative Feedback Survey of App Feasibility and Acceptability | Module 1 (approximately week 1)
  Self-report measures asking for qualitative feedback on module content and user experience.
Quantitative Feedback Survey of App Feasibility and Acceptability | Module 2 (approximately week 1)
  Self-report measures asking for qualitative feedback on module content and user experience.
Quantitative Feedback Survey of App Feasibility and Acceptability | Module 3 (approximately week 2)
  Self-report measures asking for qualitative feedback on module content and user experience.
Quantitative Feedback Survey of App Feasibility and Acceptability | Module 4 (approximately week 2)
  Self-report measures asking for qualitative feedback on module content and user experience.
Quantitative Feedback Survey of App Feasibility and Acceptability | Module 5 (approximately week 3)
  Self-report measures asking for qualitative feedback on module content and user experience.
Quantitative Feedback Survey of App Feasibility and Acceptability | Module 6 (approximately week 3)
  Self-report measures asking for qualitative feedback on module content and user experience.
Quantitative Feedback Survey of App Feasibility and Acceptability | Module 7 (approximately week 4)
  Self-report measures asking for qualitative feedback on module content and user experience.
Quantitative Feedback Survey of App Feasibility and Acceptability | Module 8 (approximately week 4)
  Self-report measures asking for qualitative feedback on module content and user experience.
Quantitative Feedback Survey of App Feasibility and Acceptability | Module 9 (approximately week 5)
  Self-report measures asking for qualitative feedback on module content and user experience.
Quantitative Feedback Survey of App Feasibility and Acceptability | Module 10 (approximately week 5)
  Self-report measures asking for qualitative feedback on module content and user experience.
Quantitative Feedback Survey of App Feasibility and Acceptability | Module 11 (approximately week 6)
  Self-report measures asking for qualitative feedback on module content and user experience.
Quantitative Feedback Survey of App Feasibility and Acceptability | Module 12 (approximately week 6)
  Self-report measures asking for qualitative feedback on module content and user experience.
Qualitative Feedback of App Feasibility and Acceptability at midpoint | Midpoint (approximately 3 weeks)
  Feedback Interviews are qualitative interview-based questionnaires that a member of the research team will lead during a phone or video call with each participant. Items will examine participant response to app content, structure, and functionality, as well as engagement and satisfaction.
Qualitative Feedback of App Feasibility and Acceptability at post-intervention | Post-intervention (approximately 6 weeks)
  Feedback Interviews are qualitative interview-based questionnaires that a member of the research team will lead during a phone or video call with each participant. Items will examine participant response to app content, structure, and functionality, as well as engagement and satisfaction.
Qualitative Feedback of App Feasibility and Acceptability at follow-up | Follow-up (approximately 12 weeks)
  Feedback Interviews are qualitative interview-based questionnaires that a member of the research team will lead during a phone or video call with each participant. Items will examine participant response to app content, structure, and functionality, as well as engagement and satisfaction.

SECONDARY OUTCOMES:
Changes in postnatal depression measures scores from baseline to midpoint as measured by the Edinburgh Postnatal Depression Scale (EPDS). | Baseline, midpoint (approximately 3 weeks)
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report measure of mood symptoms in perinatal individuals. Scores range from 0 to 30 with the following interpretation: 0-7 (depression not likely), 8-13 (depression possible), 14+ (depression probable).
Changes in postnatal depression measures scores from baseline to post-intervention as measured by the Edinburgh Postnatal Depression Scale (EPDS). | Baseline, post-intervention (approximately 6 weeks)
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report measure of mood symptoms in perinatal individuals. Scores range from 0 to 30 with the following interpretation: 0-7 (depression not likely), 8-13 (depression possible), 14+ (depression probable).
Changes in postnatal depression measures scores from midpoint to post-intervention as measured by the Edinburgh Postnatal Depression Scale (EPDS). | Midpoint (approximately 3 weeks), post-intervention (approximately 6 weeks)
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report measure of mood symptoms in perinatal individuals. Scores range from 0 to 30 with the following interpretation: 0-7 (depression not likely), 8-13 (depression possible), 14+ (depression probable).
Changes in postnatal depression measures scores from post-intervention to follow-up as measured by the Edinburgh Postnatal Depression Scale (EPDS). | Post-intervention (approximately 6 weeks), follow-up (approximately 12 weeks).
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report measure of mood symptoms in perinatal individuals. Scores range from 0 to 30 with the following interpretation: 0-7 (depression not likely), 8-13 (depression possible), 14+ (depression probable).
Changes in postnatal anxiety measures scores from baseline to midpoint as measured by the Edinburgh Postnatal Depression Scale-Anxiety Subscale (EPDS 3A). | To be completed at midpoint at approximately 3 weeks, post-intervention at approximately 6 weeks, and follow-up and approximately 12 weeks.
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report measure of mood symptoms in perinatal individuals. The Edinburgh Anxiety Subscale (EPDS 3A) uses three items from the EPDS to assess levels of anxiety among perinatal individuals. Scores range from 0 to 9, with scores of 6+ indicating likely anxiety.
Changes in postnatal anxiety measures scores from baseline to post-intervention as measured by the Edinburgh Postnatal Depression Scale-Anxiety Subscale (EPDS 3A). | Baseline, post-intervention (approximately 6 weeks)
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report measure of mood symptoms in perinatal individuals. The Edinburgh Anxiety Subscale (EPDS 3A) uses three items from the EPDS to assess levels of anxiety among perinatal individuals. Scores range from 0 to 9, with scores of 6+ indicating likely anxiety.
Changes in postnatal anxiety measures scores from midpoint to post-intervention as measured by the Edinburgh Postnatal Depression Scale-Anxiety Subscale (EPDS 3A). | Midpoint (approximately 3 weeks), post-intervention (approximately 6 weeks)
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report measure of mood symptoms in perinatal individuals. The Edinburgh Anxiety Subscale (EPDS 3A) uses three items from the EPDS to assess levels of anxiety among perinatal individuals. Scores range from 0 to 9, with scores of 6+ indicating likely anxiety.
Changes in postnatal anxiety measures scores from post-intervention to follow-up as measured by the Edinburgh Postnatal Depression Scale-Anxiety Subscale (EPDS 3A). | Post-intervention (approximately 6 weeks), follow-up (approximately 12 weeks)
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report measure of mood symptoms in perinatal individuals. The Edinburgh Anxiety Subscale (EPDS 3A) uses three items from the EPDS to assess levels of anxiety among perinatal individuals. Scores range from 0 to 9, with scores of 6+ indicating likely anxiety.
Changes in anxiety measures scores from baseline to midpoint as measured by the Generalized Anxiety Disorder-7 (GAD-7) | Baseline, midpoint (approximately 3 weeks)
  The General Anxiety Disorder-7 is a 7 item self-report measure assessing symptoms of anxiety. Scores range from 0 to 21 with the following interpretation: 0-4 (minimal anxiety), 5-9 (mild anxiety), 10-14 (moderate anxiety), 15-21 (severe anxiety).
Changes in anxiety measures scores from baseline to post-intervention as measured by the Generalized Anxiety Disorder-7 (GAD-7) | Baseline, post-intervention (approximately 6 weeks)
  The General Anxiety Disorder-7 is a 7 item self-report measure assessing symptoms of anxiety. Scores range from 0 to 21 with the following interpretation: 0-4 (minimal anxiety), 5-9 (mild anxiety), 10-14 (moderate anxiety), 15-21 (severe anxiety)
Changes in anxiety measures scores from midpoint to post-intervention as measured by the Generalized Anxiety Disorder-7 (GAD-7) | Midpoint (approximately 3 weeks), post-intervention (approximately 6 weeks)
  The General Anxiety Disorder-7 is a 7 item self-report measure assessing symptoms of anxiety. Scores range from 0 to 21 with the following interpretation: 0-4 (minimal anxiety), 5-9 (mild anxiety), 10-14 (moderate anxiety), 15-21 (severe anxiety)
Changes in anxiety measures scores from post-intervention to follow-up as measured by the Generalized Anxiety Disorder-7 (GAD-7) | Post-intervention (approximately 6 weeks), follow-up (approximately 12 weeks)
  The General Anxiety Disorder-7 is a 7 item self-report measure assessing symptoms of anxiety. Scores range from 0 to 21 with the following interpretation: 0-4 (minimal anxiety), 5-9 (mild anxiety), 10-14 (moderate anxiety), 15-21 (severe anxiety)
Change in depression measures scores from baseline to midpoint as measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline, midpoint (approximately 3 weeks)
  The PHQ-9 is a 9 item self-report measure assessing symptoms of depression. Scores range from 0 to 27 with the following interpretation: 1-4 (minimal depression), 5-9 (mild depression), 10-14 (moderate depression), 15-19 (moderately severe depression), 20-27 (severe depression).
Change in depression measures scores from baseline to post-intervention as measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline, post-intervention (approximately 6 weeks)
  The PHQ-9 is a 9 item self-report measure assessing symptoms of depression. Scores range from 0 to 27 with the following interpretation: 1-4 (minimal depression), 5-9 (mild depression), 10-14 (moderate depression), 15-19 (moderately severe depression), 20-27 (severe depression).
Change in depression measures scores from midpoint to post-intervention as measured by the Patient Health Questionnaire-9 (PHQ-9) | Midpoint, post-intervention (approximately 6 weeks)
  The PHQ-9 is a 9 item self-report measure assessing symptoms of depression. Scores range from 0 to 27 with the following interpretation: 1-4 (minimal depression), 5-9 (mild depression), 10-14 (moderate depression), 15-19 (moderately severe depression), 20-27 (severe depression).
Change in depression measures scores from post-intervention to follow-up as measured by the Patient Health Questionnaire-9 (PHQ-9) | Post-intervention (approximately 6 weeks), Follow-up (approximately 12 weeks)
  The PHQ-9 is a 9 item self-report measure assessing symptoms of depression. Scores range from 0 to 27 with the following interpretation: 1-4 (minimal depression), 5-9 (mild depression), 10-14 (moderate depression), 15-19 (moderately severe depression), 20-27 (severe depression).
Changes in perinatal trauma measure scores from baseline to post-intervention as measured by Perinatal-Post Traumatic Stress Disorder Questionnaire-II (PPQ-II) | To be completed at midpoint at approximately 3 weeks, post-intervention at approximately 6 weeks, and follow-up and approximately 12 weeks.
  The Perinatal-Post Traumatic Stress Disorder Questionnaire-II (PPQ-II) is a 14-item self-report measure assessing symptoms of trauma among postpartum individuals. Scores range from 0 to 56, with scores of 19+ distinguishing individuals in need of treatment to address symptoms.
Changes in perinatal trauma measure scores from baseline to post-intervention as measured by Perinatal-Post Traumatic Stress Disorder Questionnaire-II (PPQ-II) | Baseline, post-intervention (approximately 6 weeks)
  The Perinatal-Post Traumatic Stress Disorder Questionnaire-II (PPQ-II) is a 14-item self-report measure assessing symptoms of trauma among postpartum individuals. Scores range from 0 to 56, with scores of 19+ distinguishing individuals in need of treatment to address symptoms.
Changes in perinatal trauma measure scores from post-intervention to follow-up as measured by Perinatal-Post Traumatic Stress Disorder Questionnaire-II (PPQ-II) | Post-intervention (approximately 6 weeks), follow-up (approximately 12 weeks)
  The Perinatal-Post Traumatic Stress Disorder Questionnaire-II (PPQ-II) is a 14-item self-report measure assessing symptoms of trauma among postpartum individuals. Scores range from 0 to 56, with scores of 19+ distinguishing individuals in need of treatment to address symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Temkin-Yu, Psy.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bennett HA, Einarson A, Taddio A, Koren G, Einarson TR. Prevalence of depression during pregnancy: systematic review. Obstet Gynecol. 2004 Apr;103(4):698-709. doi: 10.1097/01.AOG.0000116689.75396.5f. PMID 15051562
- [Background] Dennis CL, Chung-Lee L. Postpartum depression help-seeking barriers and maternal treatment preferences: a qualitative systematic review. Birth. 2006 Dec;33(4):323-31. doi: 10.1111/j.1523-536X.2006.00130.x. PMID 17150072
- [Background] Furtado M, Chow CHT, Owais S, Frey BN, Van Lieshout RJ. Risk factors of new onset anxiety and anxiety exacerbation in the perinatal period: A systematic review and meta-analysis. J Affect Disord. 2018 Oct 1;238:626-635. doi: 10.1016/j.jad.2018.05.073. Epub 2018 Jun 18. PMID 29957480
- [Background] Gavin NI, Gaynes BN, Lohr KN, Meltzer-Brody S, Gartlehner G, Swinson T. Perinatal depression: a systematic review of prevalence and incidence. Obstet Gynecol. 2005 Nov;106(5 Pt 1):1071-83. doi: 10.1097/01.AOG.0000183597.31630.db. PMID 16260528
- [Background] Gaynes BN, Gavin N, Meltzer-Brody S, Lohr KN, Swinson T, Gartlehner G, Brody S, Miller WC. Perinatal depression: prevalence, screening accuracy, and screening outcomes. Evid Rep Technol Assess (Summ). 2005 Feb;(119):1-8. doi: 10.1037/e439372005-001. No abstract available. PMID 15760246
- [Background] Goodman SH, Gotlib IH. Risk for psychopathology in the children of depressed mothers: a developmental model for understanding mechanisms of transmission. Psychol Rev. 1999 Jul;106(3):458-90. doi: 10.1037/0033-295x.106.3.458. PMID 10467895
- [Background] Gjerdingen DK, Yawn BP. Postpartum depression screening: importance, methods, barriers, and recommendations for practice. J Am Board Fam Med. 2007 May-Jun;20(3):280-8. doi: 10.3122/jabfm.2007.03.060171. PMID 17478661
- [Background] Murray L. The impact of postnatal depression on infant development. J Child Psychol Psychiatry. 1992 Mar;33(3):543-61. doi: 10.1111/j.1469-7610.1992.tb00890.x. PMID 1577898
- [Background] Pearlstein T, Howard M, Salisbury A, Zlotnick C. Postpartum depression. Am J Obstet Gynecol. 2009 Apr;200(4):357-64. doi: 10.1016/j.ajog.2008.11.033. PMID 19318144
- [Background] Slomian J, Honvo G, Emonts P, Reginster JY, Bruyere O. Consequences of maternal postpartum depression: A systematic review of maternal and infant outcomes. Womens Health (Lond). 2019 Jan-Dec;15:1745506519844044. doi: 10.1177/1745506519844044. PMID 31035856
- [Background] Tietz A, Zietlow AL, Reck C. Maternal bonding in mothers with postpartum anxiety disorder: the crucial role of subclinical depressive symptoms and maternal avoidance behaviour. Arch Womens Ment Health. 2014 Oct;17(5):433-42. doi: 10.1007/s00737-014-0423-x. Epub 2014 Apr 1. PMID 24687168
- [Background] Trost SL, Beauregard JL, Smoots AN, Ko JY, Haight SC, Moore Simas TA, Byatt N, Madni SA, Goodman D. Preventing Pregnancy-Related Mental Health Deaths: Insights From 14 US Maternal Mortality Review Committees, 2008-17. Health Aff (Millwood). 2021 Oct;40(10):1551-1559. doi: 10.1377/hlthaff.2021.00615. PMID 34606354
- [Background] Wisner KL, Sit DK, McShea MC, Rizzo DM, Zoretich RA, Hughes CL, Eng HF, Luther JF, Wisniewski SR, Costantino ML, Confer AL, Moses-Kolko EL, Famy CS, Hanusa BH. Onset timing, thoughts of self-harm, and diagnoses in postpartum women with screen-positive depression findings. JAMA Psychiatry. 2013 May;70(5):490-8. doi: 10.1001/jamapsychiatry.2013.87. PMID 23487258
- [Background] Wisner KL, Hanusa BH, Perel JM, Peindl KS, Piontek CM, Sit DK, Findling RL, Moses-Kolko EL. Postpartum depression: a randomized trial of sertraline versus nortriptyline. J Clin Psychopharmacol. 2006 Aug;26(4):353-60. doi: 10.1097/01.jcp.0000227706.56870.dd. PMID 16855451
- [Derived] Temkin-Yu AB, Ayaz A, Blicker E, Liu MX, Oh A, Siegel IE, Seewald MJ, Hermann AD, Givrad S, Baez LM, Osborne LM, Green CM, Schier MM, Davis AM, Zhu S, Falk A, Bennett SM. Feasibility of a Mobile App-Based Cognitive-Behavioral Perinatal Skills Program: Protocol for Nonrandomized Pilot Trial. JMIR Res Protoc. 2025 Jan 28;14:e59461. doi: 10.2196/59461. PMID 39874578